CLINICAL TRIAL: NCT03559088
Title: Impact of Integrating a Disease-Specific Migraine App Into the Management of Patients in the Primary Care Setting
Brief Title: A Study of the Effect of a Disease-Specific Migraine Smart Phone Application (App) on Participant Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17129; I5Q-MC-CGBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine Participants Using Application (App) (Experimental): Participants with migraine history or a recent prescription for a common migraine medication will use a migraine app linked to their electronic health record (EHR) with results reported in their EHR.
  Interventions: Other: Migraine App
- Controls Not Using App (No Intervention): Observational history on contemporaneous matched controls at similar sites without migraine app linked to their EHR.

INTERVENTIONS:
Other: Migraine App — Smart phone app used to report migraine burden to the EHR.
  Arms: Migraine Participants Using Application (App)

SUMMARY:
The purpose of this study is to determine whether using a smart phone application to foster communication between study participants and their doctor will impact care. Participants must have a history of migraine or have recently been prescribed a common medicine to treat migraine. The study will last about one year for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine (ICD10: G43.*) since October 2015 OR a record of being prescribed a triptan prior to study
* Have not been prescribed a preventive migraine medication within the past twelve months
* Have not visited a neurologist in the past year
* Have an upcoming visit with their Atrium Health primary care provider

Exclusion Criteria:

* Do not own an iOS or Android smart phone with a data plan or are unwilling to install the app on their phone
* Are currently participating in a clinical trial involving an investigational drug
* Have previously used the app used in this study
* Are pregnant at the time of study entry
* Are not able to provide informed consent
* Cannot speak and read English fluently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Receiving a Preventive Migraine Prescription | Next primary care appointment following use of app (estimated as 5 weeks)
  Number of Participants Receiving a Preventive Migraine Prescription

SECONDARY OUTCOMES:
Number of Months of App Use | Baseline through one year
  Number of Months of App Use
Number of Participants Receiving Acute and Preventive Migraine Treatments, Opioids, Barbiturates | Baseline through one year
  Number of Participants Receiving Acute and Preventive Migraine Treatments, Opioids, Barbiturates
Number of Acute Care Visits | Baseline through one year
  Number of Acute Care Visits
Number of Primary Care Visits | Baseline through one year
  Number of Primary Care Visits
Number of Emergency Room Visits | Baseline through one year
  Number of Emergency Room Visits
Number of Urgent Care Visits | Baseline through one year
  Number of Urgent Care Visits
Number of Referrals to a Neurologist | Baseline through one year
  Number of Referrals to a Neurologist
Number of New Diagnoses of Migraine or Chronic Migraine | Baseline through one year
  Diagnoses made by International Classification of Diseases 10th revision (ICD10) coding system

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (16):
  - Charlotte Internal Medicine, Charlotte, North Carolina
  - Charlotte Medical Clinic, Charlotte, North Carolina
  - Carmel Family Physicians, Charlotte, North Carolina
  - Charlotte Medical Clinic-South Park, Charlotte, North Carolina
  - Randolph Internal Medicine, Charlotte, North Carolina
  - South Charlotte Primary Care, Charlotte, North Carolina
  - Mecklenburg Medical Group - Ballantyne, Charlotte, North Carolina
  - Table Rock Family Medicine, Glen Alpine, North Carolina
  - Mecklenburg Medical Group - Northcross, Huntersville, North Carolina
  - North Charlotte Medical Specialists - Huntersville, Huntersville, North Carolina
  - Lincoln Family Practice, Lincolnton, North Carolina
  - Mecklenburg Medical Group - Matthews, Matthews, North Carolina
  - Union Family Practice, Monroe, North Carolina
  - Troy Medical Services, Troy, North Carolina
  - Shiland Family Fort Mill, Fort Mill, South Carolina
  - Shiland Family Practice, Fort Mill, South Carolina